CLINICAL TRIAL: NCT06545344
Title: Preoperative, Specialty Palliative Care for Patients Considering Pancreatic Surgery: Pilot Feasibility and Acceptability Study
Brief Title: Palliative Care Consultation to Improve Communication for Patients Considering Surgery for a Pancreatic Neoplasm
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed before opening to accrual; Insufficient staff
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1124214; NCI-2024-05662 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20350 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-07-22; First posted 2024-08-09 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Usual care) (Active Comparator): Patients receive usual care and undergo evaluation by a tumor board within 14 days of baseline.
  Interventions: Other: Best Practice; Other: Survey Administration; Other: Tumor Board Review
- Arm II (Palliative care visit) (Experimental): Patients attend a palliative care visit over 60 minutes to discuss their illness, quality of life, fears and concerns and communication preferences within 7 days of baseline. Patients also undergo evaluation by a tumor board within 14 days of baseline.
  Interventions: Procedure: Palliative Care Consultation; Other: Survey Administration; Other: Tumor Board Review

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm I (Usual care)
Procedure: Palliative Care Consultation — Attend a palliative care visit
  Arms: Arm II (Palliative care visit)
Other: Survey Administration — Ancillary studies
Other: Tumor Board Review — Undergo evaluation by tumor board
  Other Names: multidisciplinary opinion

SUMMARY:
This clinical trial evaluates a palliative care consultation for improving communication between providers and patients considering surgery for a pancreatic neoplasm. Pancreatic operations have known complications that can affect quality of life. Palliative care has been shown to improve patient reported quality of life and functional outcomes. Receiving a palliative care consultation may improve communication and decision making for patients considering surgery for a pancreatic neoplasm.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive usual care and undergo evaluation by a tumor board within 14 days of baseline.

ARM II: Patients attend a palliative care visit over 60 minutes to discuss their illness, quality of life, fears and concerns and communication preferences within 7 days of baseline. Patients also undergo evaluation by a tumor board within 14 days of baseline.

After completion of study intervention, patients are followed up 7 days after the tumor board visit and 90 days after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Pancreatic neoplasm pathology
* Ability to read, write, and speak in English
* Has decisional capacity
* Expected to be seen and discussed at PCSC and seeing a surgeon as part of their tumor board evaluation

Exclusion Criteria:

* Metastatic pancreatic neoplasm
* Currently incarcerated
* Currently is or previously has received palliative care, or are unwilling to forego palliative care for the first 90 days post randomization
* Evidence of any behavior, condition, or circumstance (including, but not limited to: blindness, deafness, serious behavior or mental health conditions, discontinuing curative treatment, lack of access to technology, etc) that would interfere with their ability to complete study procedures as noted within the chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of recruited patients that consent (acceptability) | At time of consent
  Acceptability will be defined as ≥ 60% of recruited patients consented.
Percentage of patients randomized to the interventional arm who complete the palliative care consult prior to tumor board (feasibility) | At time of multidisciplinary tumor board discussion (No more than 14 days after baseline)
  Feasibility will be defined as ≥ 60% of patients randomized to interventional arm who complete palliative care consult prior to pancreatic cancer specialty clinic tumor board.

SECONDARY OUTCOMES:
Percentage of participants who complete the decisional conflict scale | At completion of 7 day follow-up timepoint
Percentage of participants who complete study measures within the first 90 days | At completion of 90 day follow-up timepoint
Percentage of participants randomized to usual care who go on to receive palliative care within the active study period | At 90 day follow-up timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Loggers, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No